CLINICAL TRIAL: NCT00618644
Title: A Phase I Study to Evaluate the Ocular and Non Ocular Safety of Ranibizumab in Treating Neovascularization Secondary to Sickle Cell Retinopathy
Brief Title: Ranibizumab for Neovascularization in Sickle Cell Retinopathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to lack of eligible participants
Sponsor: Kresge Eye Institute (Other)
Collaborators: Wayne State University (Other); Genentech, Inc. (Industry)
Responsible Party: Vinay A. Shah, M.D., Kresge Eye Institute
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 08-08; FVF4232s
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Sickle Cell Anemia; Retinopathy
MeSH Terms: conditions — Anemia, Sickle Cell; Retinal Diseases | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Ranibizumab injection
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab 0.5 mg intravitreal injection
  Other Names: Lucentis (ranibizumab)

SUMMARY:
The purpose of this study is to determine the ocular and non-ocular safety of a single dose of ranibizumab in treating neovascularization secondary to sickle cell retinopathy.

DETAILED DESCRIPTION:
In the U.S., about 10% of African Americans have an abnormal hemoglobin gene. About 8% of African Americans are heterozygous for Hemoglobin S. In the United States, sickle cell anemia primarily occurs in the black population, with approximately 0.2% of African American children afflicted by this disease. It may be associated with other hemoglobinopathies as well. The prevalence in adults is lower because of the decrease in life expectancy. Systemically, the sickle cell anemia variation (SS) produces the most symptoms. With respect to the eye, the sickle cell disease mutation (SC) produces the most effects. Overall, the sickle cell trait expression (AS) produces the fewest complications.

* Among patients with SC or SThal, the incidence of proliferation sickle cell retinopathy is 33% and 14% respectively.
* Proliferative sickle cell retinopathy is the major cause of vision loss in sickle cell disease.

For sickle cell retinopathy, the commonly used therapeutic modalities include laser retinal photocoagulation, retinal cryotherapy, and vitrectomy/membranectomy depending on the severity of the disease. The most effective therapeutic modality with minimal postoperative complications appears to be scatter laser retinal photocoagulation.

A single case study of bevacizumab was found to effective in short term regression of neovascularization and improving vision after a single injection. Further study with ranibizumab is warranted.

Recent clinical trials (Marina and Anchor) have demonstrated that ranibizumab is effective in treating patients with CNV with age-related macular degeneration. Retinopathy in sickle cell disease has also been linked to VEGF. Therefore, patients with sickle cell retinopathy should respond to ranibizumab therapy.

This is an open-label single dose, phase I study of intravitreally administered ranibizumab in patients with sickle cell retinopathy.

Consented, enrolled subjects will receive a single open-label intravitreal injection of 0.5 mg ranibizumab.

Three subjects from one site in the United States will be enrolled.

Patients will receive one dose of 0.5 mg ranibizumab administered intravitreally.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell anemia and retinopathy
* Over age 18 years
* Non-pregnant

Exclusion Criteria:

* Pregnant
* Glaucoma
* Patients using anticoagulants (e.g., warfarin)
* Retinal detachment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Ocular safety of a single dose of ranibizumab | Three months

SECONDARY OUTCOMES:
Change in vision status | Three months
To evaluate ocular hemorrhage | Three months.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Shah, MD, Principal Investigator — Kresge Eye Institute
Locations (1):
- Kresge Eye Institute, Detroit, Michigan, United States

REFERENCES:
- [Background] Al-Abdulla NA, Haddock TA, Kerrison JB, Goldberg MF. Sickle cell disease presenting with extensive peri-macular arteriolar occlusions in a nine-year-old boy. Am J Ophthalmol. 2001 Feb;131(2):275-6. doi: 10.1016/s0002-9394(00)00778-9. PMID 11228315
- [Background] McLeod DS, Merges C, Fukushima A, Goldberg MF, Lutty GA. Histopathologic features of neovascularization in sickle cell retinopathy. Am J Ophthalmol. 1997 Oct;124(4):455-72. doi: 10.1016/s0002-9394(14)70862-1. PMID 9323937
- [Background] Witkin AJ, Rogers AH, Ko TH, Fujimoto JG, Schuman JS, Duker JS. Optical coherence tomography demonstration of macular infarction in sickle cell retinopathy. Arch Ophthalmol. 2006 May;124(5):746-7. doi: 10.1001/archopht.124.5.746. No abstract available. PMID 16682603
- [Background] Chalam KV, Shah VA. Macular infarction a presentation of sickle cell crisis. Eye (Lond). 2004 Dec;18(12):1277-8. doi: 10.1038/sj.eye.6701409. No abstract available. PMID 15105819
- [Background] Avery RL. Regression of retinal and iris neovascularization after intravitreal bevacizumab (Avastin) treatment. Retina. 2006 Mar;26(3):352-4. doi: 10.1097/00006982-200603000-00016. No abstract available. PMID 16508438
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Siqueira RC, Costa RA, Scott IU, Cintra LP, Jorge R. Intravitreal bevacizumab (Avastin) injection associated with regression of retinal neovascularization caused by sickle cell retinopathy. Acta Ophthalmol Scand. 2006 Dec;84(6):834-5. doi: 10.1111/j.1600-0420.2006.00779.x. No abstract available. PMID 17083555